CLINICAL TRIAL: NCT04810585
Title: Efficacy and Biomarker Exploration of 2nd Line Aflibercept in Combination With FOLFIRI in Advanced Colorectal Cancer
Brief Title: Plasma Biomarker for Aflibercept in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1285
Record Dates: First submitted 2021-03-09; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Recurrent or Metastatic Colorectal Cancer
MeSH Terms: conditions — Recurrence; Colorectal Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Aflibercept + FOLFIRI

INTERVENTIONS:
Drug: Aflibercept + FOLFIRI — Day 1. Aflibercept + FOLFIRI
  * aflibercept(Zaltrap): 4 mg/kg IV infusion for over 1hr (Do not administer as an IV push or bolus)
  * Folinic acid: 400 mg/m2 IV infusion for over 2 hours
  * Irinotecan: 150 mg/m2 IV infusion for over 1 hours
  * 5-FU: 400 mg/m2 IV bolus injection for over 5 minute
  * 5-FU: 2400 mg/m2 IV continuous infusion for 46 hours every 2 weeks until progression disease or death or unacceptable toxicity

SUMMARY:
Based on the pervious data, aflibercept in combination with FOLFIRI is one of the effective 2nd line treatment option in advanced colorectal cancer. In this study, we prospectively assess the efficacy of 2nd line aflibercept in combination with FOLFIRI in advanced colorectal cancer in terms of progression-free survival. We further assess the efficacy according to the type of 1st line treatment. plasma biomarker study (HGF, VEGF-A, VEGF-D, IFN-γ, Angiopoietin-2, sICAM-1, sVCAM-1, TIMP-1, PIGF (HS), IL-6 (HS), IL-8 (HS), sNeuropilin-1, Thrombospondin-2 , Osteopontin , sVEGFR1, sVEGFR2, sVEGFR3) , overall survival (OS)OS, objective response rate (ORR), and safety are also assessed as the 2ndary objectives.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, single arm study. Patients will be considered "on study" upon signing the written informed consent form (ICF). The study consists of a baseline period, followed by a treatment period, consisting of 14-day treatment cycles, which will end by a 30-day Follow-up visit, which in turn, will be followed by a post-treatment follow-up period.

Patients will be evaluated for PFS then be followed on study until death or until cut-off date for final analysis of OS has been reached, whichever comes first.

During the 21-day baseline period, all baseline procedures will have to be performed within defined timelines, including review of eligibility criteria During the treatment period, the study treatment, aflibercept combined with FOLFIRI will be administered every 2 weeks unless a definitive treatment discontinuation criterion is met. Cycle lengths may be extended in case of unresolved toxicity.

Imaging to document tumor response and progressive disease will take place every 6 weeks and will continue to be done during the follow-up period in case of early study treatment discontinuation (i.e. prior to documented progression). Once disease progression is documented, patients will be followed every 2 months for survival status and collection of data regarding further anticancer therapy, until death or until the study cutoff date, whichever comes first.

The patients will be followed for safety for a minimum of 30 days following the last administration of the study treatment (30-day Follow-up visit). Beyond this date, all study drug related AEs and all SAEs should be followed until resolution/stabilization. Study drug-related AEs brought to the attention of the investigator at any time after the 30-day Follow-up visit should be recorded in the case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult, ≥ 19 years old at the time of informed consent
2. Patient has histologically confirmed advanced adenocarcinoma of colon or rectum
3. Patients who were failed in only one treatment with target agent (anti-EGFR Ab or anti-VEGF Ab) combined with FOLFOX
4. At least one measurable disease, as defined by RECIST version 1.1
5. ECOG PS of 0 to 2.
6. Life expectancy ≥ 3 months.
7. Acceptable hematologic status (without growth factor support or transfusion dependency):

   1. ANC ≧ 1.5 x 109/L,
   2. Platelet count ≧100 x 109/L
   3. Hemoglobin ≧9.0 g/dL.
8. Acceptable liver function:

   1. Bilirubin ≤ 1.0 x upper limit of normal(ULN)
   2. AST, ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN in case of liver metastasis
9. Serum creatinine ≤ 1.0 x UNL
10. Patients who understand study protocol and signed informed consents.

Exclusion Criteria:

1. Previous therapy with other VEGFR inhibitors (other than bevacizumab) or irinotecan
2. Patients who have serious underlying co-morbidities which could cause end-organ dysfunction, interfere with the conduct of the study, or that would pose an unacceptable risk to the subject in this study. in the opinion of the Investigator
3. Contraindications to the use of FOLFIRI or aflibercept
4. Female patients who are pregnant or breast feeding, or male/female patients of reproductive potential who are not willing to employ effective birth control
5. Patients who are unable to read the study consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 5years
  progressive disease (PD) or death, whichever occurs first. Results will be summarized by arm
  * Kaplan-Meier method for survival function estimate
  * Stratified Cox proportional hazard regression for hazard ratio (HR) estimate

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 5years
ORR (Objective Response Rate) | up to 5years
Incidence of Adverse events (Safety)/ vital sign(Safety)/ ECOG PS(Safety) | up to 5years
Prognostic or Predictive Biomarker for Aflibercept (plasma biomarker) | up to 5years

CONTACTS AND LOCATIONS:
Overall Officials: Joong Bae Ahn, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No